CLINICAL TRIAL: NCT04168515
Title: Lived Experiences and Impact of Delirium in Critically Ill Children: a Qualitative Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: 7280
Record Dates: First submitted 2019-09-03; First posted 2019-11-19 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient
- Caregiver
- Healthcare provider

SUMMARY:
The investigators aim to conduct a qualitative study evaluating the long and short-term recollection and experiences of critically ill children with delirium as well as collect the lived experience of the caregiver and healthcare provider involved in the patient's care. The investigators objective is to determine if there are common themes to these experiences, and if these themes are associated with specific pediatric delirium subtypes (hypoactive, hyperactive, and mixed). The overall goal is to better understand the impact of delirium on patients and their caregivers, and develop strategies to improve education, prevention and management when caring for children with pediatric intensive care unit(PICU)-acquired delirium.

DETAILED DESCRIPTION:
Summary of the project: Delirium, a disorder of brain dysfunction characterized by fluctuations in attention, consciousness and cognition, is an important but under-recognized problem in critically ill children. Well known to affect critically ill adults, we now understand that delirium also affects children, and is associated with increased mortality and length of stay as well as long-term adverse functional and quality-of-life sequelae. Delirium is common in critically ill children, affecting at least 25% of the overall population. However, the detection and management of pediatric delirium is challenging due to the lack of awareness of clinicians and researchers and the insufficient understanding of the impact delirium can have on children's physical, emotional and quality of life outcomes. Furthermore, the caregivers (family members and health care providers) of patients who witness PICU delirium will often identify their perception of the child's distress and similarly undergo their own trauma secondary to the impact of caring for the child.While there are numerous publications outlining delirium experiences in adult patients, there is no such body of research evaluating the pediatric experience. The investigators objective is to conduct a qualitative study evaluating the memories and personal experiences in critically ill children with delirium, as well as the caregiver's perception of the experience. The overall goals of this study are to build on the knowledge and understanding of PICU delirium, from the patient's perspective. To the investigator's knowledge this will be the first qualitative study on PICU delirium, and hence will be a significant contribution to this expanding field of research. These results will enable us to better understand the lived experience of delirium and thereby develop management strategies which may include modifying the PICU environment, sleep hygiene and neuro-physical rehabilitation strategies, to address this commonly acquired PICU complication and ultimately optimize the recovery of critically ill children.

Project Plan:

Aim and Objectives: The investigators aim to conduct a qualitative study evaluating the short-and long-term recollection and experiences of critically ill children with delirium. Given that a majority of children may be pre-verbal by nature of age, investigators will aim to determine the caregiver's perception of the child's experience of delirium as well as the personal impact of caring for a child with delirium. The objective is to determine if there are common themes to these experiences, and if these themes are associated with specific pediatric delirium subtypes (hypoactive, hyperactive, and mixed). The overall goal is to better understand the impact of delirium on patients and their caregivers, and develop strategies to improve education, prevention and management when caring for children with PICU-acquired delirium.

Study Design: This qualitative study will be conducted at 2 pediatric ICUs, at McMaster Children's Hospital and New York-Presbyterian Komansky Children's Hospital. The study will initially start at McMaster Children's Hospital and expand to Komansky Children's Hospital once an initial pilot study (estimated 5 interviews) is completed. Critically ill children aged under 18 years, who are diagnosed with delirium during their PICU admission, and/or their caregivers and health care providers, will be approached for consent to participate in qualitative interviews. PICU-acquired delirium will be diagnosed by the Cornell Assessment of Pediatric Delirium (CAPD) score of ≥ 9 for a duration of at least 48 hours from the PICU database. There will be 2 cohorts in the research study; 1) a retrospective cohort, having had diagnosis of delirium within the last 12 months to understand long-standing lived experience of delirium and 2) a prospective cohort with delirium diagnosis within the last 4 weeks to evaluate the immediate, short-term effects of delirium.This prospective cohort will also undergo a 2nd interview to evaluate the long-term effects of delirium.

Methods: Investigators will obtain the demographic data on each participant (age,gender, reason for PICU admission, severity of illness score (PIM 3), the details of their delirium (onset, subtype, duration and management), and which caregivers are interviewed. Hermeneutic qualitative research methods will be used in this study. Hermeneutic approaches are suitable to clarify incomplete, confusing or conflicting data, thus being a beneficial approach in qualitative research. Investigators plan to conduct face-to-face, semi-structured interviews with the patient, their family member and/or the healthcare provider involved in the care in order to understand the patient's lived experience of the event. Prospective interviews will be conducted within 4 weeks following the initial diagnosis of PICU delirium and resolution of critical illness for the child to personally participate in the interview (if cognitively able). A second interview will be conducted 2-6 months post hospital discharge, to determine if there is any perceived longer lasting impact from PICU delirium. Retrospective interviews will be conducted with patients captured from the PICU database who experienced delirium in the last 12 months while admitted to the PICU. Interviews will be guided by an interview key developed by the research team who have expertise in PICU, delirium and qualitative methods, and a patient and family member who have experienced delirium. All interviews will be audio recorded, transcribed verbatim, and anonymized. Participants will be interviewed until data saturation is reached, as is the standard of rigor in qualitative research. Investigators anticipate this will require approximately 30 patients(15 at each site).

Analysis Plan: Interview transcripts and field notes will be analyzed using inductive content analysis, whereby codes are derived directly from the data. The data will be analyzed iteratively. Three investigators, with expertise in qualitative data analysis, will independently read the transcripts in a process of open coding and by consensus, develop an initial list of codes. The initial codebook will be reviewed by all members of the research team along with the initial transcript. Inter-coder reliability will be assessed for concordance. Themes and subthemes will be derived from the data. To ensure an iterative process, the researchers will meet to discuss as a group, and agree on new themes and the addition of new codes as they emerge. NVIVO software (QSR International Pty Ltd.) will be used for data management and analysis.

Ethical consideration: This study will be conducted following institutional ethics approval and with informed consent or assent from the patient and/or family member and/or health care provider. Qualitative interviews will be conducted by trained research staff. Patient privacy will be observed,and all data will be anonymized and analyzed confidentially Expected outcomes and Impact:There is a paucity of research on what critically ill children and their caregivers experience and/or recall following a diagnosis of delirium. Current evidence suggests that clinicians do not recognize the importance or long-term impact of delirium amongst critically ill children leading to emotional, physical and quality of life morbidity. Subsequently, raising awareness, the need for routine screening, and the prevention and management of delirium are not often prioritized in many PICUs. This is the first study to the investigators knowledge, that will provide an understanding of the lived experience of delirium in children and their families within the PICU. The expected results will be important not only to clinicians who care for these children, but family members who are trying to support their children and manage their own anxieties, pediatricians who follow these patients beyond the PICU, and researchers focused on understanding survivor outcomes.

Management and Governance: The research team consists of content and methods experts in pediatric critical care, delirium, and qualitative ICU research. This bi-center study will be coordinated out of McMaster University, where the data will be managed and stored. The investigators estimate a 16-month duration to execute this study: 3 months for administrative procedures (ethics approval); 9 months for patient recruitment and completion of participant interviews at 2 sites (based on patient volume, research personnel availability, 25% delirium incidence, and 75% consent rate); an additional 4 months to complete the qualitative data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric ICU patients admitted in the last year
* less than 18 years old
* delirium during PICU admission (CAPD score equal to/greater than 9 x 48 hours)

Exclusion Criteria:

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Critically ill children aged under 18 years, who are diagnosed with delirium during their PICU admission, and/or their caregivers and health care providers, will be approached for consent to participate in qualitative interviews.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Participant lived experience of delirium based on qualitative, semi-structured interviews | 12 months
  Participants will be asked open-ended questions about their delirium experience. The interviews will be transcribed and "coded" for themes by the investigators. These codes will be input into qualitative software (NVIVO) and analyzed iteratively for each interview. As this is a qualitative study, there are no expected outcomes. Outcomes will be determined by the themes that arise from the delirium interview process.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Zetterlund P, Plos K, Bergbom I, Ringdal M. Memories from intensive care unit persist for several years--a longitudinal prospective multi-centre study. Intensive Crit Care Nurs. 2012 Jun;28(3):159-67. doi: 10.1016/j.iccn.2011.11.010. PMID 22579396
- [Background] Samuelson KA. Unpleasant and pleasant memories of intensive care in adult mechanically ventilated patients--findings from 250 interviews. Intensive Crit Care Nurs. 2011 Apr;27(2):76-84. doi: 10.1016/j.iccn.2011.01.003. Epub 2011 Mar 2. PMID 21371888
- [Background] Traube C, Silver G, Reeder RW, Doyle H, Hegel E, Wolfe HA, Schneller C, Chung MG, Dervan LA, DiGennaro JL, Buttram SD, Kudchadkar SR, Madden K, Hartman ME, deAlmeida ML, Walson K, Ista E, Baarslag MA, Salonia R, Beca J, Long D, Kawai Y, Cheifetz IM, Gelvez J, Truemper EJ, Smith RL, Peters ME, O'Meara AM, Murphy S, Bokhary A, Greenwald BM, Bell MJ. Delirium in Critically Ill Children: An International Point Prevalence Study. Crit Care Med. 2017 Apr;45(4):584-590. doi: 10.1097/CCM.0000000000002250. PMID 28079605
- [Background] Svenningsen H, Egerod I, Dreyer P. Strange and scary memories of the intensive care unit: a qualitative, longitudinal study inspired by Ricoeur's interpretation theory. J Clin Nurs. 2016 Oct;25(19-20):2807-15. doi: 10.1111/jocn.13318. Epub 2016 Jul 26. PMID 27457029
- [Background] Zhang Z, Pan L, Ni H. Impact of delirium on clinical outcome in critically ill patients: a meta-analysis. Gen Hosp Psychiatry. 2013 Mar-Apr;35(2):105-11. doi: 10.1016/j.genhosppsych.2012.11.003. Epub 2012 Dec 4. PMID 23218845
- [Background] Flaigle MC, Ascenzi J, Kudchadkar SR. Identifying Barriers to Delirium Screening and Prevention in the Pediatric ICU: Evaluation of PICU Staff Knowledge. J Pediatr Nurs. 2016 Jan-Feb;31(1):81-4. doi: 10.1016/j.pedn.2015.07.009. Epub 2015 Sep 9. PMID 26362671